CLINICAL TRIAL: NCT04860258
Title: COVID-19: A Phase 3 Multicenter Clinical Trial to Evaluate the Safety, Reactogenicity and Immunogenicity of the Investigational SARS-CoV-2 mRNA Vaccine CVnCoV in Adults 18 Years of Age and Above With Co-morbidities
Brief Title: COVID-19: A Study to Evaluate Safety, Reactogenicity and Immunogenicity of the SARS-CoV-2 mRNA Vaccine CVnCoV in Adults With Co-morbidities
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Principal Investigators and CureVac decided to terminate the trial early following a change to the risk/benefit profile.
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CV-NCOV-003; 2020-004070-22 (EudraCT Number)
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus; Covid19; SARS-CoV-2; Severe Acute Respiratory Syndrome
Keywords: Covid19; CVnCoV; SARS-CoV-2 mRNA vaccine; Vaccine; SARS; COVID; Safety; Reactogenicity; Immunogenicity
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Severe Acute Respiratory Syndrome | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CVnCoV Vaccine (Experimental): Participants will be vaccinated with CVnCoV 12 µg mRNA on Day 1 and Day 29.
  Interventions: Biological: CVnCoV Vaccine

INTERVENTIONS:
Biological: CVnCoV Vaccine — Intramuscular (IM) injection in the deltoid area, preferably in the non-dominant arm.
  Other Names: CV07050101

SUMMARY:
The primary objectives of this study are to evaluate the safety and reactogenicity profile after 1 and 2 dose administrations of investigational SARS-CoV-2 mRNA vaccine CVnCoV, and to evaluate the humoral immune responses 14 days after 2 dose administrations of CVnCoV.

DETAILED DESCRIPTION:
Study participants with the following mild to moderate per protocol defined co-morbidities will be recruited: chronic kidney disease (CKD); cardiovascular disease (CVD), chronic obstructive pulmonary disease (COPD), type-2-diabetes. After safety data review, recruitment for severe cases will be opened. No severity classification will be done for study participants with chronic human immunodeficiency virus (HIV) infection with stable aviremia 12 months prior enrollment, for renal transplant patients if stable under medication for at least 6 months prior enrollment, and for study participants with a body mass index > 32 kg/m^2.

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥18 years of age with 1 or more co-morbidities.
2. For the co-morbidities chronic kidney disease, chronic obstructive pulmonary disease (COPD), chronic cardiovascular disease and diabetes mellitus, the first 25 participants per co-morbidity should include only mild to moderate cases. Thereafter, more severe conditions may be recruited following Internal Safety Review Committee (iSRC) and Data Safety Monitoring Board (DSMB) Chair approval.
3. Participant has no overt clinical signs or symptoms of COVID-19.
4. Participant has to sign the informed consent form (ICF) before any trial procedures.
5. Participants with a life expectancy of at least 1 year as per the Investigator's assessment.
6. Expected to be compliant with protocol procedures and available for clinical follow-up through the last planned visit.
7. Physical examination without acute clinically significant findings according to the Investigator's assessment.
8. Female participants: At the time of enrollment, negative human chorionic gonadotropin (hCG) pregnancy test (serum) for women presumed to be of childbearing potential on the day of enrollment. On Day 1 (pre vaccination): negative urine pregnancy test (hCG) (only required if serum pregnancy test was performed more than 3 days before).

   Note: Women that are postmenopausal (defined as amenorrhea for ≥ 12 consecutive months prior to screening without an alternative medical cause) or permanently sterilized will be considered as not having reproductive potential.
9. Female participants of childbearing potential must use highly effective methods of birth control from 2 weeks before the first administration of the trial vaccine until 3 months following the last administration.

Exclusion Criteria:

1. A previous clinical and laboratory-confirmed diagnosis of COVID-19 within the last six months prior to screening.
2. Use of any investigational or non-registered product (vaccine or drug) other than the trial vaccine within 28 days preceding the administration of the trial vaccine, or planned use during the trial period.
3. Receipt of any other vaccines within 28 days prior to enrollment in this trial or planned receipt of any vaccine within 28 days of trial vaccine administration. Planned vaccination with an inactivated influenza vaccine is permitted.
4. Receipt of any investigational, authorized or licensed SARS-CoV-2, other coronavirus vaccine or any other lipid nanoparticles (LNP)-containing messenger ribonucleic acid vaccine prior to the administration of the trial vaccine. For authorized or licensed SARS-CoV-2: planned administration during the trial up to 6 weeks after the foreseen date of second dose administration of CVnCoV.
5. Any treatment with immunosuppressants or other immune-modifying drugs (including, but not limited to, corticosteroids, biologicals, and methotrexate) for >14 days in total within 6 months prior to the administration of the trial vaccine or planned use during the trial. For corticosteroid use, this means prednisone or equivalent, 0.5 mg/kg/day for 14 days or more. The use of inhaled, topical, or localized injections of corticosteroids (e.g., for joint pain/inflammation) is permitted.

   Note: This exclusion does not apply to the renal transplant cases and is at the Investigator's discretion for participants with other co-morbidities (e.g., COPD).
6. Participants with chronic human immunodeficiency virus (HIV) infection with controlled Hepatitis B infection with therapy or aviremic Hepatitis C may be eligible for the trial, based on the Investigator's judgment.
7. History of immune-mediated or autoimmune disease.
8. History of anaphylaxis or allergy to any component of CVnCoV or aminoglycoside antibiotics.
9. History of or current alcohol and/or drug abuse.
10. History of confirmed severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS) disease.
11. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of any dose of the trial vaccine.
12. Presence or evidence of significant uncontrolled acute or chronic medical or psychiatric illness, excluding the co-morbidities specified in the protocol. Significant medical or psychiatric illnesses include but are not limited to:

    * Uncontrolled respiratory disease.
    * Uncontrolled neurological disorders or Guillain-Barré syndrome or history of seizure, except for febrile seizures during childhood.
    * Current or past malignancy, unless completely resolved without sequelae for >5 years
13. Foreseeable non-compliance with protocol, as judged by the Investigator.
14. For female participants: pregnancy or lactation.
15. Participants with impaired coagulation or any bleeding disorder in whom an IM injection or a blood draw is contraindicated. This includes participants on treatment with anticoagulants (e.g., vitamin K antagonists, novel oral anticoagulants, and heparin). Use of platelet aggregation inhibitors is not exclusionary. However, use of anticoagulants is accepted in certain co-morbidities according to the clinical Investigator's judgment and if the international normalized ratio (INR) remains ≤3.
16. Participants employed by the Sponsor, Investigator, or trial site, or relatives of research staff working on this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - Centre Hospitalier Universitaire Saint-Pierre, Brussels
  - Université Libre de Bruxelles (ULB) - Hopital Erasme, Brussels
  - Universite Catholique de Louvain (UCL) - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Universitaire (CHU) de Liege - Domaine Universitaire du Sart Tilman, Liège

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was performed in Belgium between 22 April 2021 and 21 September 2021.
Pre-assignment Details: Of the 172 participants who were screened, 129 participants with co-morbidities known to increase the risk for (severe) COVID-19 were enrolled. Participants received investigational severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) messenger ribonucleic acid (mRNA) vaccine (CVnCoV) 12 µg on Day 1 and Day 29.
Groups:
- Chronic Kidney Disease: Participants with chronic kidney disease received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. Kidney function was ascertained from the serum creatinine measurement within the last 6 months, converted into estimated glomerular filtration rate (eGFR) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, with impaired kidney function defined as eGFR <60 mL/min/1.73m².
- Chronic Obstructive Pulmonary Disease (COPD): Participants with COPD received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. COPD included emphysema and chronic bronchitis.
- Obesity: Participants with obesity received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. Obesity was defined as a body mass index (BMI) >32 kg/m².
- Chronic Cardiovascular Disease: Participants with chronic cardiovascular disease received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. Chronic cardiovascular disease included heart failure, structural heart disorder, coronary artery disease, cardiomyopathies and arterial hypertension.
- Chronic Human Immunodeficiency Virus (HIV) Infection: Participants with chronic HIV infection received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. Participants with chronic HIV infection required stable aviremia (<50 copies/mL) and CD4 count >350/mL as documented by blood samples taken within 12 months before enrollment. Viral load <50 copies/mL over 12 months with transient changes of 50-350 copies/mL was allowed.
- Type 2 Diabetes Mellitus: Participants with type 2 diabetes mellitus received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. Participants with type 2 diabetes mellitus required diabetes mellitus to be controlled with medication [HbA1c <58 mmol/mol (7.45%)].
- Renal Transplant: Participants with renal transplant received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. Participants had a renal transplant at least a year ago under stable conditions for at least 6 months with medications, categorized as low risk of rejection.
Period: Overall Study
Arm/Group | Chronic Kidney Disease | Chronic Obstructive Pulmonary Disease (COPD) | Obesity | Chronic Cardiovascular Disease | Chronic Human Immunodeficiency Virus (HIV) Infection | Type 2 Diabetes Mellitus | Renal Transplant
Started | 1 | 1 | 52 | 33 | 33 | 7 | 2
Completed | 1 | 1 | 48 | 32 | 29 | 6 | 2
Not Completed | 0 | 0 | 4 | 1 | 4 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 1 | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) consisted of all participants who received at least 1 dose of CVnCoV and for whom any post-vaccination safety data were available.
Groups:
- Chronic Kidney Disease: Participants with chronic kidney disease received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. Kidney function was ascertained from the serum creatinine measurement within the last 6 months, converted into eGFR using the CKD-EPI equation, with impaired kidney function defined as eGFR <60 mL/min/1.73m².
- COPD: Participants with COPD received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. COPD included emphysema and chronic bronchitis.
- Obesity: Participants with obesity received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. Obesity was defined as a BMI >32 kg/m².
- Chronic HIV Infection: Participants with chronic HIV infection received SARS-CoV-2 mRNA vaccine CVnCoV 12 µg on Day 1 and Day 29. Participants with chronic HIV infection required stable aviremia (<50 copies/mL) and CD4 count >350/mL as documented by blood samples taken within 12 months before enrollment. Viral load <50 copies/mL over 12 months with transient changes of 50-350 copies/mL was allowed.
- Total: Total of all reporting groups
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant | Total
Number analyzed (Participants) | 1 | 1 | 52 | 33 | 33 | 7 | 2 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 73.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 42.7 (10.77) | 52.3 (12.36) | 43.7 (11.69) | 58.3 (9.21) | 39.0 (2.83) | 46.5 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 23 | 7 | 4 | 3 | 0 | 37
  Male | 1 | 1 | 29 | 26 | 29 | 4 | 2 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 49 | 33 | 32 | 7 | 2 | 125
  Unknown or Not Reported | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 1 | 48 | 30 | 25 | 7 | 2 | 114
  Black or African American | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 8
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 6
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Solicited Adverse Event (AE) Occurring on the Day of Vaccination and the Following 7 Days After Any Dose
Description: Reactogenicity was assessed daily via collection of solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) using paper diary cards. By definition, all solicited local AEs occurring from the time of first vaccination were considered related to trial vaccination. For solicited systemic AEs, the Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Days 29 to 36)
Population: The SAS consisted of all participants who received at least 1 dose of CVnCoV and for whom any post-vaccination safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 52 | 33 | 33 | 7 | 2
Participants
  Any solicited local AEs | 1 | 0 | 40 | 28 | 26 | 6 | 2
  Any solicited systemic AEs | 1 | 0 | 46 | 29 | 31 | 7 | 2
  Any related solicited systemic AEs | 0 | 0 | 44 | 26 | 28 | 6 | 2

2. Primary Outcome: Intensity of Solicited AEs Per US Food and Drug Administration (FDA) Toxicity Grading Scale Occurring on the Day of Vaccination and the Following 7 Days After Any Dose
Description: Reactogenicity was assessed daily via collection of solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) using paper diary cards. Intensity of solicited local AEs and solicited systemic AEs were graded per the FDA Toxicity Grading Scale at Grades 1-3, where higher grades indicate a worse outcome.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Days 29 to 36)
Population: The SAS including only participants who experienced solicited local and systemic AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 0 | 46 | 29 | 31 | 7 | 2
Participants
  Any solicited local AEs: number analyzed (Participants) | 1 | 0 | 40 | 28 | 26 | 6 | 2
  Any solicited local AEs: Grade 1 | 1 | 0 | 30 | 23 | 20 | 6 | 2
  Any solicited local AEs: Grade 2 | 0 | 0 | 9 | 4 | 6 | 0 | 0
  Any solicited local AEs: Grade 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Any solicited systemic AEs: Grade 1 | 1 | 0 | 8 | 8 | 8 | 2 | 0
  Any solicited systemic AEs: Grade 2 | 0 | 0 | 19 | 12 | 14 | 3 | 2
  Any solicited systemic AEs: Grade 3 | 0 | 0 | 19 | 9 | 9 | 2 | 0

3. Primary Outcome: Duration of Solicited AEs Occurring on the Day of Vaccination and the Following 7 Days After Any Dose
Description: Reactogenicity was assessed daily via collection of solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) using paper diary cards. Duration was calculated as consecutive days with a respective solicited AE regardless of the grade of the AE. AEs ongoing after Day 8 were included.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Days 29 to 36)
Population: The SAS including only participants who experienced solicited local and systemic AEs.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 0 | 46 | 29 | 31 | 7 | 2
days
  Any solicited local AEs: number analyzed (Participants) | 1 | 0 | 40 | 28 | 26 | 6 | 2
  Any solicited local AEs | 1.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |  | 2.2 (1.11) | 2.1 (1.21) | 2.4 (0.70) | 1.8 (0.75) | 1.0 (0.00)
  Any solicited systemic AEs | 1.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |  | 4.4 (5.06) | 4.1 (2.58) | 4.3 (3.10) | 5.4 (4.83) | 3.0 (1.41)

4. Primary Outcome: Number of Participants Who Experienced an Unsolicited AE Occurring on the Day of Vaccination and the Following 28 Days After Any Dose
Description: Diaries were used for collection of unsolicited AEs on each vaccination day and the following 28 days. In addition, participants were contacted by phone to verify whether they had any health concerns since the last visit. The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to 28 days after vaccination (Days 1 to 29 and Days 29 to 57)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 52 | 33 | 33 | 7 | 2
Participants
  Any unsolicited AEs | 1 | 1 | 27 | 14 | 19 | 4 | 1
  Any related unsolicited AEs | 1 | 1 | 12 | 5 | 7 | 1 | 1

5. Primary Outcome: Intensity of Unsolicited AEs Per the Investigator's Assessment Occurring on the Day of Vaccination and the Following 28 Days After Any Dose
Description: Diaries were used for collection of unsolicited AEs on each vaccination day and the following 28 days. In addition, participants were contacted by phone to verify whether they had any health concerns since the last visit. Participants were included only once, at the maximum severity. The Investigator made an assessment of intensity for each AE reported during the trial and assigned it to one of the following categories:
  * Mild: an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
  * Moderate: an event that caused sufficient discomfort to interfere with normal everyday activities.
  * Severe: an event that prevented normal everyday activities.
Time Frame: Up to 28 days after vaccination (Days 1 to 29 and Days 29 to 57)
Population: The SAS including only participants who experienced unsolicited AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 27 | 14 | 19 | 4 | 1
Participants
  Mild | 1 | 0 | 6 | 4 | 8 | 2 | 1
  Moderate | 0 | 1 | 17 | 7 | 10 | 1 | 0
  Severe | 0 | 0 | 4 | 3 | 1 | 1 | 0

6. Primary Outcome: Number of Participants Who Experienced a Serious Adverse Event (SAE) During the Trial
Description: An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event.
  The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to Day 57
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 52 | 33 | 33 | 7 | 2
Participants
  Any SAEs | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Any related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants Who Experienced an Adverse Event of Special Interest (AESI) During the Trial
Description: AESIs included:
  * AEs with a suspected immune-mediated etiology including potential immune-mediated diseases.
  * Other AEs relevant to SARS-CoV-2 vaccine development or the target disease.
  * Non-serious intercurrent medical conditions that may affect the immune response to vaccination was collected throughout the trial.
  Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine. The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to Day 57
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 52 | 33 | 33 | 7 | 2
Participants
  Any AESIs | 0 | 0 | 2 | 1 | 1 | 0 | 0
  Any Related AESIs | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants Seroconverting for SARS-CoV-2 Spike Protein Receptor-Binding Domain (RBD) Antibodies on Day 43
Description: Seroconversion was defined as any increase in titer in antibodies against SARS-CoV-2 RBD versus baseline. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/ authorized vaccine.
Time Frame: Baseline and Day 43
Population: The Per Protocol Immunogenicity subset (PPI) included all participants who received both doses within the windows defined in the protocol, had no major protocol deviations expected to impact the immunogenicity outcomes, had not received medical treatments (such as blood products, immunoglobulin therapy) that may interfere with any of the immunogenicity measurements and had at least 1 blood sample collected starting at 14 days (Day 43) post-second vaccination available for analysis.
Measure: Number; unit: count of seroconverted participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 38 | 21 | 18 | 5 | 2
count of seroconverted participants | 1 | 0 | 34 | 19 | 16 | 4 | 1

9. Primary Outcome: Geometric Mean Titers (GMTs) of Serum SARS-CoV-2 Spike Protein RBD Antibodies on Day 43
Description: The SARS-CoV-2 spike RBD protein-specific antibodies are expressed as GMT (geometric mean of reciprocal duplicate dilutions). Concentration/titers marked as below the lower limit of quantification (LLOQ) were arbitrary replaced by half of the LLOQ for GMT computations purpose. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Day 43
Population: The PPI included all participants who received both doses within the windows defined in the protocol, had no major protocol deviations expected to impact the immunogenicity outcomes, had not received medical treatments (such as blood products, immunoglobulin therapy) that may interfere with any of the immunogenicity measurements and had at least 1 blood sample collected starting at 14 days (Day 43) post-second vaccination available for analysis.
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 38 | 21 | 18 | 5 | 2
titers | 518.410 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 50.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 1576.121 (7.5115) | 1385.663 (5.8935) | 968.795 (4.7759) | 183.523 (2.4423) | 416.051 (20.0136)

10. Primary Outcome: Subset Participants: Number of Participants Seroconverting for SARS-CoV-2 Neutralizing Antibodies on Day 43
Description: Seroconversion was defined as any increase in titer of SARS-CoV-2 neutralizing antibodies versus baseline. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Baseline and Day 43
Population: A subset of the PPI population was included in the measurement of neutralizing activity.
Measure: Number; unit: count of seroconverted participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 23 | 11 | 11 | 5 | 2
count of seroconverted participants | 1 | 0 | 16 | 6 | 7 | 0 | 1

11. Primary Outcome: Subset Participants: GMTs of Serum SARS-CoV-2 Neutralizing Antibodies on Day 43
Description: The SARS-CoV-2 neutralizing antibodies are expressed as GMT (geometric mean of reciprocal duplicate dilutions). Concentrations/titers marked as below the LLOQ were arbitrary replaced by half of the LLOQ for GMT computations purpose. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Day 43
Population: A subset of the PPI population was included in the measurement of neutralizing activity.
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 23 | 11 | 11 | 5 | 2
titers | 14.140 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 5.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 57.426 (9.1427) | 16.042 (4.0790) | 18.778 (3.9937) | 5.000 (1.0000) | 10.000 (2.6651)

12. Secondary Outcome: Number of Participants Seroconverting for SARS-CoV-2 Spike Protein RBD Antibodies on Days 29, 120, 211 and 393
Description: as for outcome 8
Time Frame: Baseline and Days 29, 120, 211 and 393
Population: The PPI. No data was collected for Days 211 and 393 due to early study termination.
Measure: Number; unit: count of seroconverted participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 39 | 21 | 18 | 5 | 2
count of seroconverted participants
  Day 29 | 0 | 0 | 13 | 7 | 3 | 1 | 0
  Day 120: number analyzed (Participants) | 0 | 1 | 7 | 2 | 2 | 1 | 0
  Day 120 |  | 0 | 6 | 1 | 2 | 1 |
  Day 211: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 393: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: GMTs of Serum SARS-CoV-2 Spike Protein RBD Antibodies on Days 29, 120, 211 and 393
Description: The SARS-CoV-2 spike RBD protein-specific antibodies are expressed as GMT (geometric mean of reciprocal duplicate dilutions). Concentrations/titers marked as below the LLOQ were arbitrary replaced by half of the LLOQ for GMT computations purpose. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Days 29, 120, 211 and 393
Population: The PPI. No data was collected for Days 211 and 393 due to early study termination.
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 39 | 21 | 18 | 5 | 2
titers
  Day 29 | 50.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 50.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 234.464 (9.4598) | 153.351 (5.6201) | 104.230 (5.4583) | 90.306 (3.7506) | 50.000 (1.0000)
  Day 120: number analyzed (Participants) | 0 | 1 | 7 | 2 | 2 | 1 | 0
  Day 120 |  | 50.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 1861.522 (7.3966) | 179.992 (6.1193) | 174.749 (1.1589) | 554.010 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |
  Day 211: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 393: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Subset Participants: Number of Participants Seroconverting for SARS-CoV-2 Neutralizing Antibodies on Days 29 and 120
Description: as for outcome 10
Time Frame: Baseline and Days 29 and 120
Population: A subset of the PPI population was included in the measurement of neutralizing activity.
Measure: Number; unit: count of seroconverted participants
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 24 | 11 | 11 | 5 | 2
count of seroconverted participants
  Day 29 | 0 | 0 | 7 | 2 | 1 | 0 | 0
  Day 120: number analyzed (Participants) | 0 | 1 | 5 | 1 | 2 | 1 | 0
  Day 120 |  | 0 | 2 | 0 | 1 | 0 |

15. Secondary Outcome: Subset Participants: GMTs of Serum SARS-CoV-2 Neutralizing Antibodies on Days 29 and 120
Description: as for outcome 11
Time Frame: Days 29 and 120
Population: A subset of the PPI population was included in the measurement of neutralizing activity.
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
Number analyzed (Participants) | 1 | 1 | 24 | 11 | 11 | 5 | 2
titers
  Day 29 | 5.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 5.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 17.311 (7.4073) | 7.297 (2.3521) | 6.234 (2.0782) | 5.000 (1.0000) | 5.000 (1.0000)
  Day 120: number analyzed (Participants) | 0 | 1 | 5 | 1 | 2 | 1 | 0
  Day 120 |  | 5.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 26.389 (7.0380) | 5.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 7.071 (1.6325) | 5.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |

ADVERSE EVENTS:
Time Frame: Up to Day 57
Description: The SAS consisted of all participants who received at least 1 dose of CVnCoV and for whom any post-vaccination safety data were available.
Arm/Group | Chronic Kidney Disease | COPD | Obesity | Chronic Cardiovascular Disease | Chronic HIV Infection | Type 2 Diabetes Mellitus | Renal Transplant
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/52 | 0/33 | 0/33 | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/52 | 0/33 | 0/33 | 1/7 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 50/52 | 32/33 | 33/33 | 7/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Kidney Disease (N=1) | COPD (N=1) | Obesity (N=52) | Chronic Cardiovascular Disease (N=33) | Chronic HIV Infection (N=33) | Type 2 Diabetes Mellitus (N=7) | Renal Transplant (N=2)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Kidney Disease (N=1) | COPD (N=1) | Obesity (N=52) | Chronic Cardiovascular Disease (N=33) | Chronic HIV Infection (N=33) | Type 2 Diabetes Mellitus (N=7) | Renal Transplant (N=2)
Eye pain (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 26 (56) | 11 (18) | 9 (17) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 9 (11) | 6 (6) | 10 (14) | 2 (2) | 1 (2)
Chills (General disorders) | 1 (2) | 0 (0) | 24 (34) | 20 (23) | 14 (23) | 1 (1) | 1 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 44 (142) | 25 (56) | 22 (58) | 7 (15) | 2 (10)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 39 (59) | 27 (40) | 27 (41) | 6 (8) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 14 (20) | 10 (11) | 6 (8) | 2 (2) | 1 (2)
Swelling (General disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 27 (54) | 15 (31) | 9 (16) | 6 (15) | 1 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 35 (68) | 21 (39) | 19 (41) | 7 (14) | 2 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 39 (106) | 21 (44) | 21 (42) | 6 (9) | 2 (8)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 5 (6) | 4 (4) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Participant recruitment was smaller than planned due to early recruitment halt. The Principal Investigators and CureVac decided to terminate the trial early following a change to the risk/benefit profile.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT04860258/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT04860258/SAP_001.pdf